CLINICAL TRIAL: NCT02611050
Title: Treatment Decisions for Multi-vessel Coronary Artery Disease Patients
Brief Title: Treatment Decisions for Multi-vessel CAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment was not feasible
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 00028467
Record Dates: First submitted 2015-11-09; First posted 2015-11-20 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Coronary Artery Disease
Keywords: patient decision aid; multi-vessel coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Option Grid (Experimental): Patients randomized to the Option Grid arm will receive the Multi-vessel Coronary Artery Disease Option Grid at the time of enrollment. The treating physician will then discuss the patient diagnosis and treatment choice reviewing the Option Grid within the conversation to facilitate patient understanding and shared decision making
  Interventions: Behavioral: The Multi-vessel Coronary Artery Disease Option Grid
- Usual Care (Other): Patients randomized to usual care will discuss the patient diagnosis and treatment options typical to the physician's routine care.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: The Multi-vessel Coronary Artery Disease Option Grid — The Multi-vessel Coronary Artery Disease Option Grid is a patient decision aid used during the clinical visit. It is one page and contains a table a patient's frequently asked questions and the respective information for each treatment strategy. The Multi-vessel Coronary Artery Disease Option Grid was developed using patient and provider feedback and has been field-tested in clinic by cardiologists and surgeons.
  Arms: Option Grid
Behavioral: Usual Care — In usual care clinicians will discuss the patient diagnosis and treatment options typical to routine care for that clinician.
  Arms: Usual Care

SUMMARY:
This study is a multi-center randomized trial to evaluate the Multi-vessel Coronary Artery Disease Option Grid patient decision aid compared to usual care in patient reported decisional conflict, knowledge, and shared decision making.

DETAILED DESCRIPTION:
Multi-vessel coronary artery disease can be treated through percutaneous coronary intervention, coronary artery bypass grafting, or medical therapy. Treatments have risk benefit tradeoffs, making patient preference integral to the treatment decision. The Multi-vessel Coronary Artery Disease Option Grid patient decision aid was developed to improve the decision making process for patients and clinicians.

Objectives:

1. Evaluate The Multi-vessel Coronary Artery Disease Option Grid impact on patient treatment decisional conflict, knowledge, and shared decision making.

   The randomized controlled trial will compare validated and standardized measures of patient decisional conflict, shared decision making, and condition specific treatment knowledge between Option Grid and usual care patients. The investigators hypothesize Option Grid patients will have improvements in patient decisional conflict, shared decision making, and knowledge compared to usual care patients. Baseline feasibility enrollment at each site prior to randomization will be used to identify current treatment patterns, and prepare intervention delivery and fidelity. Registry data will be used to identify patient treatment received and compared between Option Grid and usual care arms.
2. Examine the physician and patient process of and factors influencing Multi-vessel Coronary Artery Disease Option Grid use.

Semi-structured interviews and process evaluations will be used to describe Option Grid use and experience and identify factors that are associated with beneficial Option Grid use.

ELIGIBILITY:
Inclusion Criteria:

* Stable multi-vessel coronary artery disease diagnosed by coronary angiography defined as left main disease (>50% stenosis) or multi-vessel coronary artery disease (>70% stenosis in two or more coronary arteries)
* At relative equipoise for at least two potential treatment options, in which the treating cardiologist or surgeon has determined the treatments are anatomically feasible and safe.

Exclusion Criteria:

* Prior coronary artery bypass grafting
* Unable to read or write English
* Not cognitively able to participate in the Option Grid as determined by clinician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-09-20 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Patient Decisional Conflict | Collected immediately following patient's Option Grid or usual care clinical discussion, usually within 15 minutes after finishing the discussion.
  The Ottawa Decisional Conflict Scale is a validated measure of a patient's feeling of conflict with the decision making experience

SECONDARY OUTCOMES:
CollaboRATE Score | Collected immediately following patient's Option Grid or usual care clinical discussion, usually within 15 minutes after finishing the discussion.
  CollaboRATE is a patient reported measure of shared decision making
Treatment Knowledge | Collected immediately following patient's Option Grid or usual care clinical discussion, usually within 15 minutes after finishing the discussion.
  Questions about multi-vessel coronary artery disease treatment knowledge. Response options are 'true/false/unsure.' Scores will be based off of the percentage of correct responses from 0 to 100
Patient Experience | Within five days of the clinical discussion
  Patient's qualitative feedback during semi-structured interviews about their decision making experience
Clinician Experience | Within five days of the clinical discussion
  Clinician's qualitative feedback during semi-structured interviews about their decision making experience
Treatment Received | Within 1 month of clinical discussion
  Identified through medical records or registry data

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth L Nichols, MS, Principal Investigator — The Dartmouth Institute
Locations (4):
- United States (4):
  - Maine Medical Center, Portland, Maine
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical Center, Albany, New York
  - Albany Stratton VA Medical Center, Albany, New York